CLINICAL TRIAL: NCT07399834
Title: Comparison of Single Tunnel Versus Double Tunnel Techniques for Coracoclavicular Stabilization in Acromioclavicular Joint Injuries, A Randomized Controlled Trial
Brief Title: Comparison of Single Tunnel Versus Double Tunnel Techniques for Coracoclavicular Stabilization in Acromioclavicular Joint Injuries
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 045/2568
Record Dates: First submitted 2026-01-20; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: AC Joint Dislocation

STUDY DESIGN:
Intervention Model Description: Patients with acute Acromioclavicular injury classified as Rockwood classification type III and above who willing to undergo the operative treatment were randomized to two groups; single tunnel group and double tunnel group
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single tunnel group (Other): Patients undergo single tunnel technique Coracoclavicular stabilization
  Interventions: Procedure: Coracoclavicular stabilization
- Double tunnel group (Other): Patients undergo double tunnel technique Coracoclavicular stabilization
  Interventions: Procedure: Coracoclavicular stabilization

INTERVENTIONS:
Procedure: Coracoclavicular stabilization — Single tunnel and double tunnel technique Coracoclavicular stabilization

SUMMARY:
The study conducted to compare both clinical and radiological outcomes comparing two techniques of Coracoclavicular-stabilization; single and double tunnel technique

DETAILED DESCRIPTION:
There are now over 150 techniques of operative treatment for Acromioclavicular joint injury. Despite no techniques used nowadays is recommended as gold standard treatment, most surgeons prefer Coracoclavicular-stabilization technique. Coracoclavicular-stabilization, providing favorable outcomes in many studies, regularly conducted with two surgical techniques which are single tunnel technique and double technique. Although, both techniques result in good biomechanic, patients underwent double tunnel technique report better clinical outcome. However, double tunnel technique compared to single tunnel technique is more challenging in surgical steps and risk intraoperative complications. This trial aims to compare both clinical and radiological outcomes of the two mentioned Coracoclavicular-stabilization techniques, in order to provide data to support treatment decision in patient with acute Acromioclavicular joint injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acute Acromioclavicular joint injury classified as Rockwood classification type III and above who willing to undergo CC-stabilization operative treatment
* Patients aged 18-45 years

Exclusion Criteria:

* Patients who had experienced shoulder surgery at the same injured shoulder side
* Patients with shoulder pathology at the same injured shoulder side
* Patients with onset of Acromioclavicular joint injury for more than 3 weeks
* Patients who decided to discontinue participating the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
ACJI score | ACJI score at preop, postop 3 months, 6 months and 1 year

SECONDARY OUTCOMES:
CC-distance difference | Measured at preop, postop 1 month, 3 months, 6 months and 1 year
  CC-distance difference measured in bilateral Zanca view

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Savang Memorial Hospital, Chon Buri, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 14. Larissa E, Philipp V, Frederik B, Management of Acute High-Grade Acromioclavicular Joint Dislocations: Comparable Clinical and Radiological Outcomes After Bidirectional Arthroscopic-Assisted Stabilization With the Single Low-Profile Suture Button Technique Versus Double-Suture Button Technique Arthroscopy. 2023;39(11):2283-2290
- [Background] 13. Jaspers M, Vueghs T, K DEM, Vundelinckx B, Ruette P, A VANR. Clavicular tunnel widening after acromioclavicular joint reconstruction: comparison between single and double clavicular tunnel techniques. Acta Orthop Belg. 2024;90(1):57-62.
- [Background] 12. Pill SG, Rush L, Arvesen J, Shanley E, Thigpen CA, Glomset JL, et al. Systematic review of the treatment of acromioclavicular joint disruption comparing number of tunnels and graft type. J Shoulder Elbow Surg. 2020;29(7S):S92-S100.
- [Background] 11. Hou Z, Graham J, Zhang Y, Strohecker K, Feldmann D, Bowen TR, et al. Comparison of single and two-tunnel techniques during open treatment of acromioclavicular joint disruption. BMC Surg. 2014;14:53.
- [Background] 10. Dumont GD, Russell RD, Knight JR, Hotchkiss WR, Pierce WA, Wilson PL, et al. Impact of tunnels and tenodesis screws on clavicle fracture: a biomechanical study of varying coracoclavicular ligament reconstruction techniques. Arthroscopy. 2013;29(10):1604-7.
- [Background] 9. Banffy MB, Uquillas C, Neumann JA, ElAttrache NS. Biomechanical Evaluation of a Single- Versus Double-Tunnel Coracoclavicular Ligament Reconstruction With Acromioclavicular Stabilization for Acromioclavicular Joint Injuries. Am J Sports Med. 2018;46(5):1070-644.
- [Background] 8. Gallagher CA, Blakeney W, Zellweger R. Acromioclavicular joint dislocation with associated brachial plexus injury. BMJ Case Rep. 2014;2014.
- [Background] 7. Arrigoni P, Brady PC, Zottarelli L, Barth J, Narbona P, Huberty D, et al. Associated lesions requiring additional surgical treatment in grade 3 acromioclavicular joint dislocations. Arthroscopy. 2014;30(1):6-10.
- [Background] 6. Tischer T, Salzmann GM, El-Azab H, Vogt S, Imhoff AB. Incidence of associated injuries with acute acromioclavicular joint dislocations types III through V. Am J Sports Med. 2009;37(1):136-9.
- [Background] 5. Chillemi C, Franceschini V, Dei Giudici L, Alibardi A, Salate Santone F, Ramos Alday LJ, et al. Epidemiology of isolated acromioclavicular joint dislocation. Emerg Med Int. 2013;2013:171609.
- [Background] 4. Kiel J, Taqi M, Kaiser K. Acromioclavicular Joint Injury. StatPearls. Treasure Island (FL) ineligible companies. Disclosure: Muhammad Taqi declares no relevant financial relationships with ineligible companies. Disclosure: Kimberly Kaiser declares no relevant financial relationships with ineligible companies.2024.
- [Background] 3. Tauber M. Management of acute acromioclavicular joint dislocations: current concepts. Arch Orthop Trauma Surg. 2013;133(7):985-95.
- [Background] 2. Fraser-Moodie JA, Shortt NL, Robinson CM. Injuries to the acromioclavicular joint. J Bone Joint Surg Br. 2008;90(6):697-707.
- [Background] 1. Berthold DP, Muench LN, Dyrna F, Mazzocca AD, Garvin P, Voss A, et al. Current concepts in acromioclavicular joint (AC) instability - a proposed treatment algorithm for acute and chronic AC-joint surgery. BMC Musculoskelet Disord. 2022;23(1):1078.